CLINICAL TRIAL: NCT07241585
Title: Vitamin D Effects on Immune Microenvironment of Nonmelanoma Skin Cancer After Photodynamic Therapy (PDT)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CASE12Z25; 5P01CA084203 (NIH)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Nonmelanoma Skin Cancer; Basal Cell Carcinoma; Squamous Cell Carcinoma
Keywords: Mohs surgery; Electrodessication & curettage; ED&C; Photodynamic therapy; PDT; Vitamin D
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell | interventions — Vitamin D; Photochemotherapy; Mohs Surgery; Curettage; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Masking only applies to Arms 2 and 3, not Arm 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1: Participants donate discarded tissue for research (No VitD/Placebo + no PDT) (Other): Participants in Arm 1 will donate discarded tissue from their scheduled standard of care Mohs surgery or ED&C. They will not be randomized to receive VitD or placebo and will not have PDT.
  Interventions: Procedure: Mohs surgery or electrodessication & curettage (ED&C) (standard of care)
- Arm 2: VitD + PDT prior to Mohs surgery or ED&C (Experimental): Participants in Arms 2 and 3 will be randomized to receive either VitD or placebo prior to PDT and Mohs surgery or ED&C visit.
  Interventions: Dietary Supplement: Vitamin D (VitD); Other: Photodynamic therapy (PDT); Procedure: Mohs surgery or electrodessication & curettage (ED&C) (standard of care)
- Arm 3: Placebo + PDT prior to Mohs surgery or ED&C (Placebo Comparator): Participants in Arms 2 and 3 will be randomized to receive either VitD or placebo prior to PDT and Mohs surgery or ED&C visit.
  Interventions: Other: Placebo; Other: Photodynamic therapy (PDT); Procedure: Mohs surgery or electrodessication & curettage (ED&C) (standard of care)

INTERVENTIONS:
Dietary Supplement: Vitamin D (VitD) — Participants will orally take 10,000 international units daily of VitD for the 6 days prior to their scheduled PDT visit. Participants in Arms 2 and 3 will be blinded to whether they are receiving VitD or placebo.
  Arms: Arm 2: VitD + PDT prior to Mohs surgery or ED&C
Other: Placebo — Participants will orally take a placebo (gelatin) capsule for the 6 days prior to their scheduled PDT visit. Participants in Arms 2 and 3 will be blinded to whether they are receiving VitD or placebo.
  Arms: Arm 3: Placebo + PDT prior to Mohs surgery or ED&C
Other: Photodynamic therapy (PDT) — PDT involves a topical photosensitizing agent called aminolevulinate (ALA) being applied to the tumor surface. ALA is then activated by shining a blue light on the skin, causing a photodynamic reaction to occur. Participants will receive PDT 1-14 days prior to their scheduled Mohs surgery or ED&C visit.
  Arms: Arm 2: VitD + PDT prior to Mohs surgery or ED&C; Arm 3: Placebo + PDT prior to Mohs surgery or ED&C
Procedure: Mohs surgery or electrodessication & curettage (ED&C) (standard of care) — Participants are eligible for this study by already planning to undergo Mohs surgery or ED&C, which will be conducted per standard of care. For Arms 2 and 3, participants will undergo Mohs surgery or ED&C 1-14 days after their PDT visit. For Arm 1, participants will undergo Mohs surgery or ED&C at their scheduled time. All participants donate their discarded tissue from the Mohs surgery for research.

SUMMARY:
This research study is for people who have been diagnosed with a nonmelanoma skin cancer (either basal cell carcinoma or squamous cell carcinoma) and are planning to receive either Mohs surgery or ED&C (electrodessication & curettage) as part of clinical care. The purpose of this study is to understand how photodynamic therapy (PDT) with or without Vitamin D can promote an immune response to skin cancer.

For this study, participants will be randomized (randomly assigned) and asked to take Vitamin D or placebo for 6 days and come to the clinic for a single PDT treatment 1-14 days prior to their surgery. At this visit, photographs of participant's skin cancer will be taken, and participants will undergo PDT treatment. The study team will also take photos on the day of Mohs surgery or ED&C. There will be up to two blood draws for research.

If participants do not want to come in for a PDT treatment prior to their Mohs surgery or ED&C, they will have the option to participate by only allowing the study team to collect data about their skin cancer and their tissue from Mohs surgery or ED&C.

DETAILED DESCRIPTION:
This research study explores the effect of photodynamic therapy (PDT) on nonmelanoma skin cancers (NMSC). NMSC are made up of basal cell carcinoma (BCC) and squamous cell carcinoma (SCC). PDT is a treatment for NMSC that may be used instead of surgery. PDT uses light and a special chemical reaction to kill cancer cells on the skin's surface. First, an agent called aminolevulinate (ALA) is put on the skin of the tumor. Then, a bright blue light is shined on the skin, which causes a chemical reaction to occur. This chemical reaction helps to damage and kill cancer cells.

NMSCs are common and can usually be cured with surgery. However, surgery can leave scars or result in disfigurement. This can be especially difficult for people who have tumors on their face or other visible or sensitive parts of the body. As an alternative to surgery, photodynamic therapy (PDT) is approved in Europe to treat BCC and SCC. However, because PDT does not work as well on thicker tumors, the U.S. FDA has not yet approved it for use on NMSC in this country. Investigators want to better understand how PDT damages and kills tumor cells, so that knowledge can be used to make the treatment more effective.

Vitamin D (VitD) is both a nutrient and a steroid-like hormone. Over 10+ years of research in investigators' laboratory has shown that VitD works well with PDT to treat NMSC. When participants receive a high dose of VitD before PDT, the treatment is able to clear the tumor more effectively. This has been shown in studies with mice that had early skin cancer, as well as mice with thick skin cancer. It has also been shown to be effective in participants with BCC. One reason that VitD may help is because it increases the amount of photosensitizing agent that can accumulate within the tumor, which helps to effectively kill cancer cells with PDT when light is applied. However, VitD has another important effect, which is that it helps to attract immune cells into the tumor. This effect has been seen in mouse models of SCC. The primary purpose of this study is to further investigate this immune mechanism in humans.

ELIGIBILITY:
Inclusion Criteria:

* Must be an adult participant (> 18 yrs) who is scheduled to undergo Mohs surgery or ED&C within the Dermatologic Surgery unit of the Department of Dermatology, Cleveland Clinic.
* Must have at least one BCC or SCC tumor eligible for removal by Mohs surgery.
* The original tumor size prior to biopsy must be >1.0 cm (in the longest diameter).
* Participants of any ethnic group are eligible for this trial.
* Must provide informed consent to participate in the trial.
* Participant must live in Ohio (Groups 2 & 3), because Research Pharmacy cannot ship the study drugs outside of the state.

Exclusion Criteria:

* Pregnant or breastfeeding
* Currently being treated for other cancers with medical or radiation therapy
* Known hypersensitivity to 5-aminolevulinic acid
* History of a photosensitivity disease, e.g., porphyria cutanea tarda

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Expression of immune checkpoint molecules | At time of Mohs surgery or ED&C, up to Day 20
  Expression of immune checkpoint molecules will be compared in tumors and peri-tumoral stroma after photodynamic therapy (PDT) versus tumors without PDT and is defined as changes in the expression of PD-1, PD-L1, and TIM3, among other checkpoint inhibitors. This will be measured using the scRNA-seq data obtained from tumor tissues via Parse Biosciences scRNA-seq analysis.

SECONDARY OUTCOMES:
Ratio of cytotoxic T cells to regulatory T cells | At time of Mohs surgery or ED&C, up to Day 20
  Ratio of cytotoxic T cells to regulatory T cells will be compared in tumors and peri-tumoral stroma after photodynamic therapy (PDT) versus tumors without PDT. This is measured using scRNA-seq data (Parse Bioscienes scRNA-sequencing kit).
Ratio of M1 macrophages to M2 macrophages | At time of Mohs surgery or ED&C, up to Day 20
  Ratio of M1 macrophages to M2 macrophages will be compared in tumors and peri-tumoral stroma after photodynamic therapy (PDT) versus tumors without PDT. This is measured using scRNA-seq data (Parse Bioscienes scRNA-sequencing kit).
Proportion of tumor-activated CD8+ T-cells in circulating T-cells | At time of Mohs surgery or ED&C, up to Day 20
  Proportion of tumor-activated CD8+ T-cells in circulating T-cells will be compared in tumors and peri-tumoral stroma after photodynamic therapy (PDT) versus tumors without PDT. This will be measured using peripheral blood analyzed using fluorescence-labelling and flow analysis (FACS)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Maytin, MD, PhD, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication
Access Criteria: Request to the PI

REFERENCES:
- [Background] Braathen LR, Szeimies RM, Basset-Seguin N, Bissonnette R, Foley P, Pariser D, Roelandts R, Wennberg AM, Morton CA; International Society for Photodynamic Therapy in Dermatology. Guidelines on the use of photodynamic therapy for nonmelanoma skin cancer: an international consensus. International Society for Photodynamic Therapy in Dermatology, 2005. J Am Acad Dermatol. 2007 Jan;56(1):125-43. doi: 10.1016/j.jaad.2006.06.006. PMID 17190630
- [Background] Pogue BW, Chen B, Ochoa MI, Petusseau A, Liu A, Gibson ALF, Maytin EV, Wilson BC. Emerging uses of 5-aminolevulinic-acid-induced protoporphyrin IX in medicine: a review of multifaceted, ubiquitous, molecular diagnostic, therapeutic, and theranostic opportunities. J Biomed Opt. 2025 Dec;30(Suppl 3):S34112. doi: 10.1117/1.JBO.30.S3.S34112. Epub 2025 Oct 8. PMID 41070141
- [Background] Ortenzio MP, Anand S, Travers JB, Maytin EV, Rohan CA. Immunomodulatory effects of photodynamic therapy for skin cancer: Potential strategies to improve treatment efficacy and tolerability. Photochem Photobiol. 2025 Jul 4. doi: 10.1111/php.70008. Online ahead of print. PMID 40616218
- [Background] Anand S, Shen A, Cheng CE, Chen J, Powers J, Rayman P, Diaz M, Hasan T, Maytin EV. Combination of vitamin D and photodynamic therapy enhances immune responses in murine models of squamous cell skin cancer. Photodiagnosis Photodyn Ther. 2024 Feb;45:103983. doi: 10.1016/j.pdpdt.2024.103983. Epub 2024 Jan 27. PMID 38281610
- [Background] Maytin EV, Hasan T. Vitamin D and Other Differentiation-promoting Agents as Neoadjuvants for Photodynamic Therapy of Cancer. Photochem Photobiol. 2020 May;96(3):529-538. doi: 10.1111/php.13230. Epub 2020 Apr 15. PMID 32077114
- [Background] Anand S, Wilson C, Hasan T, Maytin EV. Vitamin D3 enhances the apoptotic response of epithelial tumors to aminolevulinate-based photodynamic therapy. Cancer Res. 2011 Sep 15;71(18):6040-50. doi: 10.1158/0008-5472.CAN-11-0805. Epub 2011 Aug 1. PMID 21807844
- [Background] Bullock TA, Mack JA, Negrey J, Kaw U, Hu B, Anand S, Hasan T, Warren CB, Maytin EV. Significant Association of Poly-A and Fok1 Polymorphic Alleles of the Vitamin D Receptor with Vitamin D Serum Levels and Incidence of Squamous Cutaneous Neoplasia. J Invest Dermatol. 2023 Aug;143(8):1538-1547. doi: 10.1016/j.jid.2023.01.028. Epub 2023 Feb 20. PMID 36813159
- [Background] Maytin EV, Zeitouni NC, Updyke A, Negrey JT, Shen AS, Heusinkveld LE, Mack JA, Hu B, Anand S, Maytin TA, Giostra L, Bullock T, Warren CB, Hasan T. High-dose oral vitamin D in combination with photodynamic therapy can accelerate the clearance rate of basal cell carcinoma: A randomized clinical trial. Photodiagnosis Photodyn Ther. 2025 Oct;55:104704. doi: 10.1016/j.pdpdt.2025.104704. Epub 2025 Jul 7. PMID 40633744
- [Background] Anand S, Hasan T, Maytin EV. Treatment of nonmelanoma skin cancer with pro-differentiation agents and photodynamic therapy: Preclinical and clinical studies (Review). Photochem Photobiol. 2024 Nov-Dec;100(6):1541-1560. doi: 10.1111/php.13914. Epub 2024 Feb 4. PMID 38310633